CLINICAL TRIAL: NCT03034772
Title: A Randomized Controlled Trial Comparing the Effect of Topical Dorzolamide-Timolol Versus Placebo Combined With Intravitreal Anti-Vascular Endothelial Growth Factor (VEGF) Injections in Patients With Neovascular Age-Related Macular Degeneration Who Are Incomplete Anti-VEGF Responders
Brief Title: Dorzolamide-timolol in Combination With Anti-vascular Endothelial Growth Factor Injections for Wet Age-related Macular Degeneration
Acronym: DAWN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Jason Hsu, MD, Co-director of Retina Research, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-596
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Neovascular Age-related Macular Degeneration; Wet Macular Degeneration
Keywords: neovascular; wet; age-related; macular degeneration; dorzolamide; timolol
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration | interventions — dorzolamide-timolol combination; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dorzolamide-timolol (Active Comparator): Topical dorzolamide-timolol twice daily for the study duration. All patients will continue to receive intravitreal anti-VEGF injections at regularly scheduled intervals.
  Interventions: Drug: Dorzolamide-timolol
- Artificial tears (Placebo Comparator): Topical artificial tears twice daily for the study duration. All patients will continue to receive intravitreal anti-VEGF injections at regularly scheduled intervals.
  Interventions: Other: Artificial tears

INTERVENTIONS:
Drug: Dorzolamide-timolol — Topical eye drop (active comparator) used twice daily for study duration
  Other Names: Cosopt
  Arms: Dorzolamide-timolol
Other: Artificial tears — Topical eye drop (placebo comparator) used twice daily for study duration
  Arms: Artificial tears

SUMMARY:
A previous pilot study demonstrated that commonly available glaucoma drops (dorzolamide-timolol) might decrease the amount of chronic swelling in patient with wet age-related macular degeneration who have been receiving anti-vascular endothelial growth factor (VEGF) injections. This will be a larger study where subjects are randomly assigned to receive the glaucoma drops or a placebo (artificial tears) in order to confirm whether this previous finding is valid. Subjects will continue to receive the normally scheduled anti-VEGF injections at regular intervals as done prior to enrollment. The only addition to the regimen will be the daily use of eye drops (dorzolamide-timolol or artificial tears) twice daily for the duration of the study. At the end of the study, the swelling in the retina will be compared to the amount before starting the drops to see if there is any difference between the group using dorzolamide-timolol versus artificial tears.

DETAILED DESCRIPTION:
Intravitreal anti-vascular endothelial growth factor (VEGF) agents, including ranibizumab and aflibercept, remain the standard of care treatment for neovascular age-related macular degeneration (AMD). Various treatment modalities using these agents have been proposed, including monthly, pro re nata, and treat-and-extend regimens. Despite frequent and consistent treatment with anti-VEGF therapy, there is a subset of patients who are incomplete responders and have persistent exudation, including intraretinal edema, subretinal fluid (SRF), and/or retinal pigment epithelial detachment (PED) on spectral-domain optical coherence tomography (SD-OCT). While clearance of intravitreal anti-VEGF drugs is not completely understood, some studies have suggested that outflow through the anterior chamber may play a role. We hypothesized that by decreasing aqueous production, outflow may also be reduced which could subsequently slow the clearance of intravitreal drugs. In a prior pilot study with 10 eyes of 10 patients who were incomplete responders with neovascular AMD, the effect of topical dorzolamide-timolol in combination with continued intravitreal anti-VEGF injections was explored. Patients were kept on the same anti-VEGF drug as well as the same interval between injections for the 2 visits before enrollment and through the course of the pilot study in order to minimize the chances that any changes noted might be the result of altering one of these variables. The mean central subfield thickness (CST) decreased from 419.7 μm at enrollment to 334.1 μm at the final visit (p=0.012). Mean maximum subretinal fluid (SRF) height decreased from 126.6 μm at enrollment to 56.5 μm at the final visit (p=0.020). This decrease in mean CST and SRF was significant beginning at the first visit after initiation of the drops. Based on this initial pilot data, dorzolamide-timolol appears to be a promising adjuvant treatment in combination with anti-VEGF injections for incomplete anti-VEGF responders with neovascular AMD. However, since there was no control group in the pilot study, it is possible that the decreased exudation seen was a result of the continued anti-VEGF therapy alone rather than an effect of the topical therapy. As a result, a randomized, placebo-controlled clinical trial will be better able to assess the efficacy of dorzolamide-timolol in this setting.

ELIGIBILITY:
Inclusion Criteria:

1. Active choroidal neovascularization (CNV) due to AMD.
2. Prior treatment with at least 4 injections of anti-VEGF agents in the past 6 months and persistent intraretinal and/or subretinal fluid on SD-OCT at each visit during this period.
3. Baseline CST ≥ 270 µm on SD-OCT automated retinal thickness map.
4. Injection of the same anti-VEGF agent at each of the two visits immediately preceding study enrollment.
5. Time interval of 5 weeks (± 1 week) between visits for at least two visits immediately preceding study enrollment.
6. Subjects of either gender aged ≥ 45 years.
7. Provide written informed consent
8. Ability to comply with study and follow-up procedures and return for study visits.

Exclusion Criteria:

1. History of uveitis.
2. Presence of intraocular inflammation, significant epiretinal membrane (causing distortion of macular anatomy per investigator discretion), significant vitreomacular traction (per investigator discretion), macular hole, or vitreous hemorrhage.
3. Any ophthalmic surgery within previous 6 months, including cataract extraction.
4. Any history of vitrectomy or glaucoma surgery (e.g., trabeculectomy, tube shunt).
5. Current prescription eye drop usage (e.g., glaucoma drops, corticosteroid drops, etc.).
6. Any contraindication for topical use of a beta-blocker (e.g., bradycardia, decompensated heart failure, chronic obstructive pulmonary disease, reactive airway disease, asthma, etc.).
7. Any history of sulfonamide allergy.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye
Locations (5):
- United States (5):
  - Palo Alto Medical Foundation, Palo Alto, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania
  - Retina Consultants of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sridhar J, Hsu J, Shahlaee A, Garg SJ, Spirn MJ, Fineman MS, Vander J. Topical Dorzolamide-Timolol With Intravitreous Anti-Vascular Endothelial Growth Factor for Neovascular Age-Related Macular Degeneration. JAMA Ophthalmol. 2016 Apr;134(4):437-43. doi: 10.1001/jamaophthalmol.2016.0045. PMID 26914218
- [Derived] Hsu J, Patel SN, Wolfe JD, Shah CP, Chen E, Jenkins TL, Wibbelsman TD, Obeid A, Mikhail M, Garg SJ, Ho AC, Chiang A, Spirn MJ, Vander JF. Effect of Adjuvant Topical Dorzolamide-Timolol vs Placebo in Neovascular Age-Related Macular Degeneration: A Randomized Clinical Trial. JAMA Ophthalmol. 2020 May 1;138(5):560-567. doi: 10.1001/jamaophthalmol.2020.0724. PMID 32239190

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Since multiple centers were enrolling simultaneously, two more patients then anticipated were randomized
Period: Overall Study
Arm/Group | Dorzolamide-timolol | Artificial Tears
Started | 27 | 25
Completed | 27 | 23
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dorzolamide-timolol | Artificial Tears | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.7 (7.5) | 77.5 (6.3) | 78.4 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 23 | 50
Intravitreal anti-vascular endothelial growth factor agent used [Count of Participants; unit: Participants]
  Aflibercept | 13 | 14 | 27
  Ranibizumab | 14 | 9 | 23
Number of prior anti-vascular endothelial growth factor (VEGF) injections [Mean (Standard Deviation); unit: injections] | 20 (15.6) | 21.1 (11.6) | 20.5 (14)
Injection interval before enrollment [Count of Participants; unit: Participants]
  Every 4 weeks | 17 | 12 | 29
  Every 5 weeks | 3 | 8 | 11
  Every 6 weeks | 7 | 3 | 10
Visual Acuity (logarithm of the minimum angle of resolution, logMAR) [Mean (Standard Deviation); unit: logMAR] | 0.37 (0.31) | 0.348 (0.19) | 0.361 (0.26)
Intraocular Pressure [Mean (Standard Deviation); unit: mm Hg] | 14.37 (2.9) | 14.22 (3.1) | 14.3 (2.95)
Baseline Optical Coherence Tomography (OCT) Measurements [Mean (Standard Deviation); unit: microns]
  Central subfield thickness | 348.3 (75.5) | 321.3 (80.5) | 335.9 (78.2)
  Maximum pigment epithelial detachment height | 230.2 (116.4) | 178.9 (111) | 206.1 (115.7)
  Maximum subretinal fluid height | 103.15 (68.5) | 90 (70.5) | 96.98 (69.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Central Subfield Thickness (CST)
Description: Change in mean CST on spectral domain optical coherence tomography from baseline to the final visit
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Dorzolamide-timolol | Artificial Tears
Number analyzed (Participants) | 27 | 23
microns | -36.6 (54) | 1.7 (52.3)
Statistical Analysis 1: Comparison: Dorzolamide-timolol vs Artificial Tears; Test type: Superiority; p = 0.04, ANCOVA; Mean difference between the 2 groups derived using analysis of covariance, with the baseline value and type of anti-VEGF drug used as covariates

2. Secondary Outcome: Change in Mean Maximum Subretinal Fluid (SRF) Height
Description: Change in mean maximum SRF height on spectral domain optical coherence tomography from baseline to final visit.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Dorzolamide-timolol | Artificial Tears
Number analyzed (Participants) | 27 | 23
microns | -49.4 (55) | -22.2 (56)
Statistical Analysis 1: Comparison: Dorzolamide-timolol vs Artificial Tears; Test type: Superiority; p = 0.11, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Mean Maximum Pigment Epithelial Detachment (PED) Height
Description: Change in mean maximum PED height on spectral domain optical coherence tomography from baseline to final visit.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Dorzolamide-timolol | Artificial Tears
Number analyzed (Participants) | 27 | 23
microns | -39.1 (65) | 1.1 (16)
Statistical Analysis 1: Comparison: Dorzolamide-timolol vs Artificial Tears; Test type: Superiority; p = 0.01, ANCOVA; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Visual Acuity
Description: Change in mean best available visual acuity from baseline to final visit.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Dorzolamide-timolol | Artificial Tears
Number analyzed (Participants) | 27 | 23
logMAR | 0.031 (0.15) | 0.018 (0.16)
Statistical Analysis 1: Comparison: Dorzolamide-timolol vs Artificial Tears; Test type: Superiority; p = 0.78, ANCOVA

5. Secondary Outcome: Change in Mean Intraocular Pressure (IOP)
Description: Change in mean IOP from baseline to final visit.
Time Frame: Baseline and 18 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dorzolamide-timolol | Artificial Tears
Number analyzed (Participants) | 27 | 23
mm Hg | -1.81 (3.8) | -0.78 (2.8)
Statistical Analysis 1: Comparison: Dorzolamide-timolol vs Artificial Tears; Test type: Superiority; p = 0.24, ANCOVA

ADVERSE EVENTS:
Time Frame: 20 months
Arm/Group | Dorzolamide-timolol | Artificial Tears
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dorzolamide-timolol (N=27) | Artificial Tears (N=25)
Eyelid edema (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03034772/Prot_SAP_001.pdf